CLINICAL TRIAL: NCT02228343
Title: A Prospective Trial of Ayurveda for Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Robert DuBroff, Principal Investigator, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNM2013.1
Record Dates: First submitted 2014-08-21; First posted 2014-08-29 (Estimated); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Medicine, Ayurvedic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ayurveda (Experimental): Ayurvedic therapy
  Interventions: Other: Ayurveda

INTERVENTIONS:
Other: Ayurveda — Ayurveda includes meditation, yoga, breathing exercises, herbs

SUMMARY:
Can Ayurvedic therapy improve markers of cardiovascular health and cardiovascular risk factors in patients with coronary artery disease.

DETAILED DESCRIPTION:
Patients with established coronary artery disease will be treated with 90 days of Ayurvedic therapy to include yoga, meditation, breathing exercises,and herbs. Arterial stiffness, weight, BMI, BP, medications, cholesterol, LDL, HDL, triglyceride, HS-CRP will be measured at baseline and after 90 days of therapy.

ELIGIBILITY:
Inclusion Criteria:

* stable coronary artery disease (prior mi, coronary angioplasty or stent, coronary bypass surgery)

Exclusion Criteria:

* age < 18 years
* life expectancy < 6 months
* pregnancy or breast feeding
* unwilling or unable to complete 90 days of therapy
* already receiving/taking Ayurvedic therapy
* unable to converse in or understand English language

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J DuBroff, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Medical Group McMahon Cardiology, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ayurveda
Started | 22
Completed | 19
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ayurveda
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not collected
  Male | NA — Data not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Participants With Arterial Stiffness Were Measured as Pulse Wave Velocity Meters/Second
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ayurveda
Number analyzed (Participants) | 19
Participants | 19

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ayurveda
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes